CLINICAL TRIAL: NCT04307966
Title: Addressing the Double Burden of Diseases Through a Pre-adolescent Transdisciplinary Intervention for Inter-generational Outcomes
Brief Title: Effectiveness of a Pre-adolescent Inter-generational Intervention to Address HIV and Obesity
Status: Completed | Type: Observational
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: Fogarty Clinical Research Inc. (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Keshni Arthur, Mrs, University of Witwatersrand, South Africa
Other Study IDs: UWitwatersrand
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Hiv; Obesity
Keywords: inter-generational outcomes; Pre-adolescents
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: 537 pre-adolescent grade 6 learners and their parent (n=537) were invited to participate. Trained educators delivered lessons about HIV and obesity to all Grade 6 students at 5 government-run schools. The classroom curriculum for students required delivery of a five-hour face-to-face intervention delivered weekly through 10 30-minute lessons. Students were asked to communicate their learnings to their parents at home. Parents were requested to read through the lesson in a workbook and to sign acknowledgement that they had read the content. The workbook contained shared student-parent homework activities that took approximately 30 minutes per week. Data was only collected from Learners (n=425) and parents (n= 427)who had consented to the study. A pretest was conducted. The intervention was then implemented. A posttest was conducted afterwards. Both parents and learners answered self-reported questionnaires.
  Interventions: Behavioral: The CIrCLE of Life Initiative

INTERVENTIONS:
Behavioral: The CIrCLE of Life Initiative — HIV and obesity prevention programme delivered directly to Grade 6 preadolescents and indirectly to their parents.

SUMMARY:
The study evaluates an intervention, The CIrCLE of Life Initiative, which was developed to address HIV and obesity prevention. We evaluated whether the combined HIV and obesity intervention increased knowledge, enhanced skills, and/or promoted healthy behaviour among pre-adolescent students (9-12 years old) and their parents.

DETAILED DESCRIPTION:
The CIrCLE of Life Initiative had both a school and home component, each comprising a learning curriculum, environmental support, and activity-based constituents that aimed to increase student knowledge and skills, and to engage parents. Trained educators delivered lessons about HIV and obesity to all Grade 6 students at 5 government-run schools. The classroom curriculum for students required delivery of a five-hour face-to-face intervention delivered weekly through 10 30-minute lessons. Students were asked to communicate their learnings to their parents at home. Parents were requested to read through the lesson in a workbook and to sign acknowledgement that they had read the content. The workbook contained shared student-parent homework activities that took approximately 30 minutes per week.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Ages: 9 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: All Grade 6 learners and their parents from 5 government-run primary schools
Sampling Method: Non-Probability Sample
Enrollment: 852 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
HIV/AIDS-related knowledge, attitude, behaviour, practices and skills | 3 months
  The primary outcome was the effects and differences between the student, pretest and posttest, and the parent, pretest and posttest.
obesity-related awareness, attitude and skills | 3 months
  The primary outcome was the effects and differences between the student, pretest and posttest, and the parent, pretest and posttest.
nutrition-related awareness, attitude, behaviour and skills | 3 months
  The primary outcome was the effects and differences between the student, pretest and posttest, and the parent, pretest and posttest.
physical activity-related awareness, attitude, behaviour and skills | 3 months
  The primary outcome was the effects and differences between the student, pretest and posttest, and the parent, pretest and posttest.
child-parent communication | 3 months
  The primary outcome was the effects and differences between the student, pretest and posttest, and the parent, pretest and posttest.

SECONDARY OUTCOMES:
pre-adolescent parent inter-generational knowledge transfer | 3 months
  The second outcome determined whether the intervention, delivered to students, could influence knowledge transfer and translation in parents.

CONTACTS AND LOCATIONS:
Overall Officials: Gill Nelson, PHD, Study Director — University of the Witwatersrand, South Africa; Nicola Christofides, PHD, Study Director — University of the Witwatersrand, South Africa
Locations (5):
- South Africa (5):
  - Kamogelo Primary school, Westonaria, Gauteng
  - Westonaria primary school, Westonaria, Gauteng
  - Westonaria primary mine school, Westonaria, Gauteng
  - Zuurbekom Primary School, Westonaria, Gauteng
  - Izanokhanyo Primary school, Westonaria, Gauteng

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: CSR
Time Frame: Data has already been made available.
URL: https://zenodo.org/record/3679352#.XmlHeC2B3LY

REFERENCES:
- [Derived] Arthur K, Christofides N, Nelson G. Effectiveness of a pre-adolescent inter-generational intervention to address HIV and obesity in South Africa, using a pretest-posttest design. BMC Public Health. 2021 Dec 11;21(1):2251. doi: 10.1186/s12889-021-12228-z. PMID 34895196